CLINICAL TRIAL: NCT07155655
Title: Influence of Motivation Combined With Motor Imagery or Action Observation on Lumbo-Pelvic Strength in Asymptomatic Subjects: A Pilot Randomised Controlled Trial
Brief Title: Influence of Motivation and Mental Practice on Lumbo-Pelvic Strength in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mateo Riera Marco (Other)
Responsible Party: Sponsor-Investigator, Mateo Riera Marco, Independent Researcher _ Sponsor-Investigator, MarcoMateoRiera
Organization: MarcoMateoRiera (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMR2023PilotRCT
Record Dates: First submitted 2025-08-19; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers; Muscle Strength
Keywords: Motor imagery; Action observation; Motivation; Lumbo-pelvic strength; Pilot trial.

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Motor Imagery (MI) (Experimental): Ten asymptomatic participants assigned to a motor imagery training protocol, performed twice weekly for four weeks.
  Interventions: Behavioral: Motor Imagery (MI)
- Action Observation (AO) (Experimental): Ten asymptomatic participants assigned to an action observation training protocol, performed twice weekly for four weeks.
  Interventions: Behavioral: Action Observation (AO)
- Motor Imagery With Motivation (MIm) (Experimental): Ten asymptomatic participants assigned to motor imagery training combined with a motivational protocol, performed twice weekly for four weeks.
  Interventions: Behavioral: Motor Imagery with Motivation (MIm)
- Action Observation With Motivation (AOm) (Experimental): Ten asymptomatic participants assigned to action observation training combined with a motivational protocol, performed twice weekly for four weeks.
  Interventions: Behavioral: Action Observation with Motivation (AOm)

INTERVENTIONS:
Behavioral: Motor Imagery (MI) — Participants followed an audio-guided motor imagery protocol describing the lumbopelvic dynamometer movement. The audio was played three times per session, with pauses for visualization. Training was delivered online via Microsoft Teams, twice weekly for four weeks, in a quiet and focused environment.
  Other Names: Mental imagery
  Arms: Motor Imagery (MI)
Behavioral: Action Observation (AO) — Participants viewed three videos of the lumbopelvic dynamometer movement (two third-person, one first-person perspective). Each video was watched three times per session. Training was delivered online via Microsoft Teams, twice weekly for four weeks, with participants instructed to remain silent and focused.
  Other Names: Observation training
  Arms: Action Observation (AO)
Behavioral: Motor Imagery with Motivation (MIm) — Participants followed the MI protocol, combined with a motivational strategy. Intrinsic motivation was provided through self-talk statements, and extrinsic motivation through an audio simulating a weightlifting competition. Each motivational audio was played three times per session. Training was delivered online via Microsoft Teams, twice weekly for four weeks.
  Arms: Motor Imagery With Motivation (MIm)
Behavioral: Action Observation with Motivation (AOm) — Participants followed the AO protocol, combined with the same motivational strategy described for the MIm group (self-talk + extrinsic audio simulation). Each motivational audio was played three times per session. Training was delivered online via Microsoft Teams, twice weekly for four weeks.
  Arms: Action Observation With Motivation (AOm)

SUMMARY:
This pilot randomized controlled trial investigated the influence of motivation combined with motor imagery (MI) or action observation (AO) on lumbo-pelvic strength in asymptomatic adults. The purpose was to explore whether adding a motivational protocol to mental practice strategies could enhance strength outcomes.

Forty healthy participants were randomly assigned to one of four groups: motor imagery (MI), action observation (AO), motor imagery with motivation (MIm), or action observation with motivation (AOm). Lumbo-pelvic strength was measured using a dynamometer, while imagery ability was evaluated with the revised Movement Imagery Questionnaire (MIQ-R). Assessments were performed at baseline and post-intervention, with strength additionally measured pre-, intra-, and post-intervention.

The trial was conducted between September 2022 and June 2023 at Centro de Estudios Universitarios La Salle, Madrid, Spain, during the investigator's student affiliation. This study is being registered retrospectively to meet ethical and publication requirements.

DETAILED DESCRIPTION:
Mental practice strategies such as motor imagery (MI) and action observation (AO) are increasingly applied in both sports and rehabilitation contexts to enhance motor learning, strength, and functional outcomes. These techniques activate neural circuits that overlap with those involved in actual movement execution and have been shown to produce both neurophysiological and performance-related changes. Motivation, an important factor in motor performance, may further influence the effectiveness of MI and AO, but its specific contribution remains unclear.

This pilot randomized controlled trial was designed to provide preliminary evidence regarding the effect of motivation combined with MI or AO on lumbo-pelvic strength in asymptomatic adults. The trial included 40 participants randomly assigned to one of four groups: MI, AO, MI with motivation, and AO with motivation. Interventions were delivered online over four weeks, with strength and imagery ability assessed at multiple time points.

The study was conducted at Centro de Estudios Universitarios La Salle (Madrid, Spain) between September 2022 and June 2023. This record is submitted retrospectively to comply with ethical and publication requirements.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic male and female participants
* Aged between 18 and 65 years
* No musculoskeletal, systemic, neurological, cognitive, or psychological disorders affecting the lumbopelvic area

Exclusion Criteria:

* Students enrolled in bioscience-related degrees beyond their first year
* History of pathology or surgery involving the lower limb or lumbar spine
* Lumbopelvic or lower limb pain within the past three months
* Illiteracy
* Pregnant women or those who suspected pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-18 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
Lumbo-pelvic strength | Baseline (Day 1), Mid-intervention (Week 2), and Post-intervention (Week 4, end of program)
  Maximal voluntary contraction of lumbo-pelvic muscles assessed using a dynamometer. Strength was recorded at three time points: baseline, mid-intervention (fourth teletraining session, Week 2), and post-intervention (Week 4, end of program).

SECONDARY OUTCOMES:
Fear of Movement | Baseline and post-intervention (4 weeks)
  Assessed using the Spanish 11-item version of the Tampa Scale for Kinesiophobia (TSK-11), which has demonstrated good reliability and validity. The scale distinguishes between two factors: Activity Avoidance and Harm. It shows strong internal consistency (Cronbach's α = 0.78) and test-retest reliability (0.81). Total scores range from 11 to 44, with higher scores indicating greater perceived kinesiophobia.
Physical activity | Baseline and post-intervention (4 weeks)
  Measured using the Spanish validated version of the International Physical Activity Questionnaire - Short Form (IPAQ-SF). This tool classifies individuals into low, moderate, and vigorous physical activity levels. The short IPAQ has shown moderate reliability (r = 0.76; 95% CI: 0.73-0.77).
Self-Efficacy for Physical Activity | Baseline and post-intervention (4 weeks)
  Assessed with a validated and reliable self-efficacy scale for physical activity (Cronbach's α > 0.9; β = 0.96). The scale includes three factors:
  * Adherence to structured exercise (three or more sessions of at least 20 minutes per week; 23 items).
  * Daily physical activity self-efficacy (13 items).
  * Daily walking self-efficacy, including perceived barriers to walking 60, 90, or 120 minutes per day (3 items).
Motor Imagery Ability - Visual and Kinaesthetic | Baseline and post-intervention (4 weeks)
  Assessed using the revised Movement Imagery Questionnaire (MIQ-R), an 8-item self-report inventory with two subscales (visual and kinaesthetic). Internal consistency is high (Cronbach's α > 0.84 for the full scale; 0.80 for visual; 0.84 for kinaesthetic). Each item involves whole-body, upper limb, or lower limb movements. The assessment includes four steps: (1) a posture is described and assumed, (2) a movement is described and performed, (3) the subject returns to the starting position and imagines performing the movement without moving, and (4) they rate how easily they could visualise or feel the imagined movement. Time to complete each imagined action is also recorded. A 7-point Likert scale is used, with "1" = very difficult to see/feel and "7" = very easy to see/feel.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Universitario La Salle - Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided